CLINICAL TRIAL: NCT03044431
Title: Autologous Stem Cell Treatment for Chronic Lung Disease Study
Status: Completed | Type: Observational
Sponsor: Lung Institute (Industry)
Responsible Party: Principal Investigator, Melissa Rubio, PhD, APRN, PhD, APRN, Lung Institute
Other Study IDs: LI001
Record Dates: First submitted 2017-02-03; First posted 2017-02-07 (Estimated); Results first posted 2017-10-25 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: COPD; Interstitial Lung Disease
Keywords: Shortness of breath; Breathlessness; Stem cells; Platelet rich plasma; Quality of life; Pulmonary Function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial; Dyspnea | interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cell therapy treated: All patients/participants enrolled will undergo cell therapy
  Interventions: Procedure: Cell therapy

INTERVENTIONS:
Procedure: Cell therapy — Each participant will receive cell therapy with stem cells harvested either from peripheral blood or from bone marrow plus peripheral blood; after harvest, cells are processed and returned to the patient via peripheral circulation on the same day.

SUMMARY:
The purpose of the Lung Institute is to collect and isolate a patient's own cells and platelet rich plasma (PRP) and deliver the product back to the patient the same day. Lung Institute's treatment is limited to self-funded patients with chronic lung disease- chronic obstructive pulmonary disease (COPD) and restrictive lung diseases such as pulmonary fibrosis (PF) and interstitial lung disease (ILD). The patient's cells and platelet rich plasma are harvested through venous or bone marrow collection techniques.

The hypothesized outcomes of therapy are safety and minimization of adverse events, a perceived improvement in the patient's lung condition (to be determined by their perceived quality of life), an improvement in the FEV1 among COPD patients, the ability to reduce supplemental oxygen use, the ability to function well without the use of rescue inhalers, reduction of secondary pulmonary infections, reduction in emergency room visits and exacerbations related to their disease.

DETAILED DESCRIPTION:
Through the collection of outcomes data, Lung Institute aims to explore and describe the safety and efficacy of autologous stem cell treatment for chronic lung disease with dissemination to the public and to the medical community for the advancement of regenerative medicine. The study aims to confirm the safety of autologous cell therapy, explore the effect of autologous cell therapy treatment on pulmonary function over time, and to describe the anecdotal quality of life changes of patients following treatment using quantitative and qualitative measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients are included in treatment by self-referral and after consultation with a designated patient coordinator who determines initial eligibility, and then by the clinic nurse practitioner or physician of Lung Institute who determines final eligibility for inclusion. All eligible treated patients are eligible for the study.

Exclusion Criteria:

* Patients who are unable to provide informed consent, pregnant patients, prisoners, non-English speakers, patients with a history of cancer within the past 5 years, patients with active tuberculosis or pneumonia. In addition, patients on prescribed blood thinners, with a history of breast or prostate cancer of any time frame or with a history of osteoporosis are excluded from the bone marrow harvest option.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include all patients treated with cell therapy Lung Institute in Dallas, Texas.
Sampling Method: Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Rubio, PhD, APRN, Principal Investigator — Lung Institute Dallas
Locations (1):
- Lung Institute Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinic webpage — http://lunginstitute.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients who underwent elective, investigational cell therapy were enrolled in the outcomes study.
Pre-assignment Details: No patients in the study received placebo. All patients received autologous, adult stem cell therapy.
Period: Overall Study
Arm/Group | Cell Therapy Treated
Started | 207
Completed | 148
Not Completed | 59
Not completed — Lost to Follow-up | 59

BASELINE CHARACTERISTICS:
Population: All patients who underwent cell therapy were included in the data analysis.
Arm/Group | Cell Therapy Treated
Number analyzed (Participants) | 207
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 165
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95
  Male | 112
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Number of Participants with Chronic Obstructive Pulmonary Disease (COPD) [Count of Participants; unit: Participants] | 167
Number of Participants with Interstitial Lung Disease (ILD) [Count of Participants; unit: Participants] | 40
Treatment Type [Count of Participants; unit: Participants]
  Venous Protocol | 159
  Double Venous Protocol | 26
  Bone Marrow Protocol | 22
Baseline FEV1 if participant has COPD [Mean (Full Range); unit: FEV1 Percentage (%)] — Population: 167 patients in the overall sample were diagnosed with chronic obstructive pulmonary disease (COPD).
  FEV1 Percentage (%)
    number analyzed (Participants) | 167
    (all) | 36.9 [9 to 85]
Baseline Clinical COPD Questionnaire Score All Participants [Mean (Full Range); unit: units on a scale] — The Clinical COPD Questionnaire (CCQ) is a 10-item scale where the participant chooses responses on a 0-6 scale for each item. 0 represents no symptoms and 6 represents severe symptoms. The mean of the responses is the final score and ranges from 0-6, 0 is least severe symptoms and 6 is most severe symptoms.
  units on a scale | 3.6 [0.8 to 6.0]
COPD Participant Baseline QOL (quality of life) score based on the Clinical COPD Questionnaire (CCQ) [Mean (Full Range); unit: units on a scale] — The Clinical COPD Questionnaire (CCQ) is a 10-item scale where the participant chooses responses on a 0-6 scale for each item. 0 represents no symptoms and 6 represents severe symptoms. The mean of the responses is the final score and ranges from 0-6, 0 is least severe symptoms and 6 is most severe symptoms. Population: 167 patients in the overall sample had a diagnosis of COPD.
  units on a scale
    number analyzed (Participants) | 167
    (all) | 3.6 [1.0 to 6.0]
ILD Participant Baseline QOL score based on Clinical COPD Questionnaire (CCQ) [Mean (Inter-Quartile Range); unit: units on a scale] — The Clinical COPD Questionnaire (CCQ) is a 10-item scale where the participant chooses responses on a 0-6 scale for each item. 0 represents no symptoms and 6 represents severe symptoms. The mean of the responses is the final score and ranges from 0-6, 0 is least severe symptoms and 6 is most severe symptoms. Population: 40 patients in the sample were diagnosed with interstitial lung disease (ILD)
  units on a scale
    number analyzed (Participants) | 40
    (all) | 3.3 [0.8 to 5.6]

OUTCOME MEASURES:

1. Primary Outcome: Change in FEV1 From Baseline Among COPD Patients
Description: Change from baseline (among COPD patients only) as measured by pulmonary function testing/spirometry at baseline and again at 6 months post- treatment
Time Frame: Measurements pre-treatment and then at 6 months post- treatment
Population: All patients with COPD were asked to provide a 6 month post-treatment pulmonary function test. 5 participants completed and returned the test.
Measure: Mean (Full Range); unit: percentage of change in FEV1
Arm/Group | Cell Therapy Treated
Number analyzed (Participants) | 5
percentage of change in FEV1 | 12.8 [0 to 100]

2. Primary Outcome: Number of Participants Reporting an Improvement in 3 Month-Post Treatment QOL Scores, All Diagnoses
Description: Number of patients in the total sample who reported an improved perceived quality of life 3 months post-treatment as measured by the Clinical COPD Questionnaire (CCQ).
Time Frame: Measurements pre-treatment and then at 3 months post-treatment for all diagnoses
Population: 148 of 207 enrolled participants completed the 3 month post-treatment QOL survey
Measure: Count of Participants; unit: Participants
Arm/Group | Cell Therapy Treated
Number analyzed (Participants) | 148
Participants | 121

3. Primary Outcome: Number of Participants Reporting an Improvement in 6 Month-Post Treatment QOL Scores, All Diagnoses
Description: Number of patients in the total sample who reported an improved perceived quality of life 6 months post-treatment as measured by the Clinical COPD Questionnaire (CCQ).
Time Frame: Measurements pre-treatment and then at 6 months post-treatment among all diagnoses
Population: 124 patients completed a 6 month post-treatment QOL survey
Measure: Count of Participants; unit: Participants
Arm/Group | Cell Therapy Treated
Number analyzed (Participants) | 124
Participants | 90

4. Other Pre Specified Outcome: Number of Participants With COPD Reporting an Improvement in 3 Month-Post Treatment QOL Scores
Description: Number of patients with a diagnosis of COPD who reported an improved perceived quality of life 3 months post-treatment as measured by the Clinical COPD Questionnaire (CCQ).
Time Frame: Measurements for COPD pre-treatment and then at 3 months post-treatment
Population: 120 patients with COPD completed a 3 month post-treatment QOL survey
Measure: Count of Participants; unit: Participants
Arm/Group | Cell Therapy Treated
Number analyzed (Participants) | 120
Participants | 102

5. Other Pre Specified Outcome: Number of Participants With COPD Reporting an Improvement in 6 Month-Post Treatment QOL Scores
Description: Number of patients with a diagnosis of COPD who reported an improved perceived quality of life 6 months post-treatment as measured by the Clinical COPD Questionnaire (CCQ).
Time Frame: Measurements for COPD pre-treatment and then at 6 months post-treatment
Population: 101 patients with COPD completed a 6 month post-treatment QOL survey
Measure: Count of Participants; unit: Participants
Arm/Group | Cell Therapy Treated
Number analyzed (Participants) | 101
Participants | 79

6. Other Pre Specified Outcome: Number of Participants With Interstitial Lung Disease Reporting an Improvement in 3 Month-Post Treatment QOL Scores
Description: Number of patients with a diagnosis of Interstitial Lung Disease who reported an improved perceived quality of life 3 months post-treatment as measured by the Clinical COPD Questionnaire (CCQ).
Time Frame: Measurements for ILD pre-treatment and then at 3 months post-treatment
Population: 28 patients with ILD completed a 3 month post-treatment QOL survey
Measure: Count of Participants; unit: Participants
Arm/Group | Cell Therapy Treated
Number analyzed (Participants) | 28
Participants | 20

7. Other Pre Specified Outcome: Number of Participants With Interstitial Lung Disease Reporting an Improvement in 6 Month-Post Treatment QOL Scores
Description: Number of patients with a diagnosis of Interstitial Lung Disease who reported an improved perceived quality of life 6 months post-treatment as measured by the Clinical COPD Questionnaire (CCQ).
Time Frame: Measurements for ILD pre-treatment and then at 6 months post-treatment
Population: 23 patients with ILD completed a 6 month post-treatment QOL survey
Measure: Count of Participants; unit: Participants
Arm/Group | Cell Therapy Treated
Number analyzed (Participants) | 23
Participants | 13

ADVERSE EVENTS:
Time Frame: Adverse events monitoring and reporting was done over the entire length of the study, approximately 11 months from March 2016 through December 2016.
Description: Any and all adverse events were reported to the Principal Investigator and reported to MaGil IRB and the supporting organization's quality and compliance monitor within 48 hours of the event.
Arm/Group | Cell Therapy Treated
All-Cause Mortality (participants affected / at risk) | 4/207
Serious Adverse Events (participants affected / at risk) | 0/207
Other Adverse Events (participants affected / at risk) | 10/207
OTHER ADVERSE EVENTS (reported when occurring in more than 0.2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cell Therapy Treated (N=207)
Dizziness (Surgical and medical procedures) | 7 (7) — Participant reported dizziness following collection of blood sample for venous cell therapy.
Bradycardia, not procedure related (Cardiac disorders) | 1 (1) — Participant presented with pre-treatment significant bradycardia and was transported to the emergency department for evaluation. Treatment protocol stopped pending evaluation.
Hypotension (Cardiac disorders) | 2 (2) — Participants experienced low blood pressure following bone marrow harvesting of stem cells. Blood pressure was immediately corrected by the participant laying down and receiving intravenous fluids.

LIMITATIONS AND CAVEATS:
This study is limited by a small sample size for post-treatment pulmonary function test returns and the self-reporting of quality of life scores. The CCQ measure quantifiable and can show trends over time, but it remains a subjective measure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-09-22): https://cdn.clinicaltrials.gov/large-docs/31/NCT03044431/Prot_SAP_ICF_000.pdf